CLINICAL TRIAL: NCT00238368
Title: Autologous Blood or Marrow Transplantation for Aggressive Non-Hodgkin's Lymphoma Based on Early [18F] FDG-PET Scanning
Brief Title: Fludeoxyglucose F 18 Positron Emission Tomography in Predicting Risk of Relapse in Patients With Non-Hodgkin's Lymphoma Who Are Undergoing Combination Chemotherapy With or Without Autologous Stem Cell or Bone Marrow Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Diagnostic
Other Study IDs: J0348 CDR0000445618; P30CA006973 (NIH); JHOC-J0348; JHOC-03082605
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Lymphoma
Keywords: contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage I adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; contiguous stage II grade 3 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; stage I grade 3 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 3 follicular lymphoma; anaplastic large cell lymphoma; stage I adult T-cell leukemia/lymphoma; stage II adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Large-Cell, Anaplastic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Filgrastim; Rituximab; Busulfan; Cisplatin; Cyclophosphamide; Cytarabine; Doxorubicin; Etoposide; Methylprednisolone; Prednisone; Vincristine; Peripheral Blood Stem Cell Transplantation; Magnetic Resonance Spectroscopy; Fluorodeoxyglucose F18; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Biological: rituximab
Drug: busulfan
Drug: cisplatin
Drug: cyclophosphamide
Drug: cytarabine
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: methylprednisolone
Drug: prednisone
Drug: vincristine sulfate
Procedure: autologous bone marrow transplantation
Procedure: peripheral blood stem cell transplantation
Procedure: positron emission tomography
Radiation: fludeoxyglucose F 18
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells. Giving chemotherapy with an autologous stem cell or bone marrow transplant may allow more chemotherapy to be given so that more cancer cells are killed. Procedures, such as fludeoxyglucose F 18 positron emission tomography (FDG-PET) (done during chemotherapy) may help doctors predict a patient's risk of relapse and help plan the best treatment.

PURPOSE: This phase II trial is studying how well FDG-PET works in predicting risk of relapse in patients with aggressive non-Hodgkin's lymphoma who are undergoing combination chemotherapy with or without autologous stem cell or bone marrow transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine event-free survival of patients with aggressive non-Hodgkin's lymphoma treated with early high-dose therapy and autologous peripheral blood stem cell (PBSC) or bone marrow transplantation (BMT) based on positive fludeoxyglucose F 18 positron emission tomography (FDG-PET) results obtained during first-line chemotherapy.
* Compare event-free survival of patients treated with this regimen with historical event-free survival of patients with positive FDG-PET results obtained during first-line chemotherapy that are not treated with early high-dose therapy.

Secondary

* Compare overall survival of patients treated with a standard treatment regimen vs early high-dose therapy and autologous PBSC or BMT based on FDG-PET results obtained during first-line chemotherapy.
* Determine the predictive value of an early negative FDG-PET result in these patients.
* Correlate International Prognostic Index risk category with FDG-PET results and overall outcome in these patients.

OUTLINE: This is a pilot study.

* First-line chemotherapy: Patients receive cyclophosphamide IV, doxorubicin IV, and vincristine IV on day 1, oral prednisone on days 1-5, and rituximab IV on day 1 (patients with CD20-positive disease only) OR another standard first-line chemotherapy regimen. Treatment repeats every 14-21 days for 2 or 3 courses in the absence of disease progression or unacceptable toxicity.
* Radiographic staging: Between days 11-20 of course 2 or 3 OR days 11-13 of course 3 of first-line chemotherapy, patients receive fludeoxyglucose F 18 (FDG) IV. One hour later, patients undergo whole-body FDG-positron emission tomography (PET) and CT scan. Patients with no evidence of malignant disease by FDG-PET (i.e., negative result) receive a standard treatment regimen that may include localized radiotherapy for limited stage or bulky disease followed, 4-6 weeks later, by a repeat whole-body FDG-PET and CT scan. Patients with progressive disease after first-line chemotherapy are removed from the study. Patients with evidence of malignant disease by FDG-PET (i.e., positive result) and stable disease or better proceed to ESHAP chemotherapy.
* ESHAP chemotherapy: Patients receive etoposide IV over 2 hours, methylprednisolone IV, and cisplatin IV over 3 hours on days 1-4 followed by cytarabine IV over 2 hours on day 5. Patients with CD20-positive disease also receive rituximab IV on day 1. Treatment repeats every 14-21 days for 2 courses in the absence of disease progression or unacceptable toxicity. Beginning 1 day after completion of course 2, patients receive filgrastim (G-CSF) subcutaneously once daily followed by leukapheresis to collect peripheral blood stem cells (PBSC). Some patients may also undergo bone marrow (BM) harvest if sufficient PBSC are not collected. Patients with a sufficient number of stem cells proceed to high-dose therapy and autologous PBSC transplantation (PBSCT) or BM transplantation (BMT).
* High-dose therapy and PBSCT or BMT: No more than 4 weeks after completion of PBSC collection or BM harvest, patients receive high-dose therapy that may include cyclophosphamide and total-body irradiation OR busulfan and cyclophosphamide. Patients then undergo PBSCT or BMT. Between 4-6 weeks after completion of PBSCT or BMT, patients undergo repeat whole-body FDG-PET and CT scan. Patients may also undergo consolidative radiotherapy to the sites of bulky disease at the discretion of the physician.

After completion of study treatment, patients are followed at 4 weeks, every 3 months for 2 years, every 6 months for 1 year, and then annually for 2 years.

PROJECTED ACCRUAL: A total of 55 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed aggressive non-Hodgkin's lymphoma of 1 of the following subtypes:

  * Diffuse large B-cell lymphoma
  * Mediastinal (thymic) B-cell lymphoma
  * Grade 3 follicular lymphoma
  * Anaplastic large cell lymphoma
  * Peripheral T-cell lymphoma
* Must have adequate staging of disease by the following techniques:

  * CT scan or MRI of affected sites
  * Bone marrow biopsy (in cases where results influence the duration of chemotherapy only)
  * Lumbar puncture (if clinically indicated)
* Stage I-IV disease
* Any International Prognostic Index risk category
* Radiographically measurable disease
* None of the following aggressive non-Hodgkin's subtypes are allowed:

  * Mantle cell lymphoma
  * Lymphoblastic lymphoma
  * Burkitt's lymphoma
  * Mycosis fungoides/Sezary's syndrome
  * HTLV-1-associated T-cell leukemia/lymphoma
  * Primary CNS lymphoma
  * HIV-associated lymphoma
  * Transformed lymphomas
* No prior diagnosis of another hematologic malignancy
* No known progressive disease during prior first-line chemotherapy
* No active CNS involvement by lymphoma, except CNS involvement at diagnosis that is previously treated and in remission

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-4 (0-2 for peripheral blood stem cell [PBSC] or bone marrow transplantation [BMT] patients)

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count > 1,000/mm^3*
* Platelet count ≥ 75,000/mm^3 NOTE: *PBSC or BMT patients only

Hepatic

* Bilirubin ≤ 2.0 mg/dL unless due to Gilbert's disease or lymphoma*
* No known significant hepatic dysfunction that is not expected to improve and would preclude PBSC or BMT NOTE: *PBSC or BMT patients only

Renal

* Creatinine ≤ 2.0 mg/dL*
* No known significant renal dysfunction that is not expected to improve and would preclude PBSC or BMT NOTE: *PBSC or BMT patients only

Cardiovascular

* Ejection fraction ≥ 45% by echocardiogram or MUGA*
* No known significant cardiac dysfunction that is not expected to improve and would preclude PBSC or BMT NOTE: *PBSC or BMT patients only; a cardiology consult and evaluation may override ejection fraction criterion

Pulmonary

* FEV_1 and FVC ≥ 50% of predicted for patients who have not received thoracic or mantle radiotherapy (75% of predicted for patients who have received thoracic or mantle radiotherapy)*
* No known significant pulmonary dysfunction that is not expected to improve and would preclude PBSC or BMT NOTE: *PBSC or BMT patients only

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 3 years except carcinoma in situ of the cervix or nonmelanoma skin cancer
* No known HIV positivity OR HIV negative (for PBSC or BMT patients only)
* No serious illness that would preclude study participation
* No contraindication to autologous BMT

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* No more than 3 prior courses of chemotherapy for lymphoma

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2004-02 (Actual); Primary Completion 2007-09-17 (Actual); Study Completion 2007-09-17 (Actual)

PRIMARY OUTCOMES:
2-year event free survival

SECONDARY OUTCOMES:
Overall survival
Predictive value of early negative fludeoxyglucose F 18 positron emission tomography (FDG-PET)
Correlation of International Prognostic Index risk category with FDG-PET results and overall outcome

CONTACTS AND LOCATIONS:
Overall Officials: Lode J. Swinnen, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States